CLINICAL TRIAL: NCT05522127
Title: A Comparison of Restrictive and Liberal Fluid Administration During Elective Colonoscopy Under Sedoanalgesia
Brief Title: Restritive and Liberal Fluid Management and Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yonca Özvardar Pekcan, MD, Anesthesia and Reanimation specialist, principal investigator, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KA22/87
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Intravenous Infusions; Colonoscopy; Sedoanalgesia
Keywords: Sedoanalgesia; Colonoscopy; Intravenous Infusions
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Restrictive) (Active Comparator): Group R (Restrictive, 2ml/kg 0.9% NaCl during colonoscopy)
  Interventions: Other: Colonoscopy; Other: Sedoanalgesia
- Group L (Liberal ) (Active Comparator): Group L (Liberal 15ml/kg 0.9% NaCl during colonoscopy)
  Interventions: Other: Colonoscopy; Other: Sedoanalgesia

INTERVENTIONS:
Other: Colonoscopy — Colonoscopy
Other: Sedoanalgesia — Ketamine, fentanil, midazolam, propofol

SUMMARY:
intraduction and aim In this study, in cases who will undergo elective day colonoscopy under sedoanalgesia; It was planned to investigate the effects of restrictive and liberal fluid administration on hemodynamics, side effects, drug levels, patient satisfaction, recovery and discharge times during the procedure.

Methods This study was planned to be conducted as a prospective, randomized (closed envelope method), controlled, double-blind study with 100 adult patients aged 18-65 years in the american sociological association (ASA I-II) risk group who will undergo colonoscopy under sedation-analgesia under elective conditions.Vascular access will be opened and randomly divided into two groups as Group R (Restrictive, 2ml/kg 0.9% Sodium cloride-NaCl during colonoscopy) and Group L (Liberal 15ml/kg 0.9% NaCl during colonoscopy). For sedoanalgesia, Midazolam 0.02 mg/kg, Fentanyl 1 μg/kg, Ketamine 0.3 mg/kg will be administered intravenous (IV), followed by 10 mg additional doses of propofol until the Ramsay sedation score (RSS) is 3-4. All colonoscopy procedures will be performed by the same gastroenterologist.

Expectations and scientific contributions This research may help to understand the effects of giving or not administering intravenous fluids (restrictive/liberal) prior to the procedure in patients undergoing elective colonoscopy under sedoanalgesia. It can provide hemodynamic stability, reduction in drug doses, reduction of side effects, rapid recovery and discharge, and reduction of costs.

DETAILED DESCRIPTION:
intraduction and aim Intestinal cleansing and restriction of oral fluid intake in preparation for colonoscopy, which is one of the most frequently performed diagnostic procedures, may cause adverse hemodynamic effects during the procedure. These adverse effects can be prevented by intravenous fluid therapy. In this study, in cases who will undergo elective day colonoscopy under sedoanalgesia; It was planned to investigate the effects of restrictive and liberal fluid administration on hemodynamics, side effects, drug levels, patient satisfaction, recovery and discharge times during the procedure.

Methods This study was planned to be conducted as a prospective, randomized (closed envelope method), controlled, double-blind study with 100 adult patients aged 18-65 years in the american sociological association (ASA) I-II risk group who will undergo colonoscopy under sedation-analgesia under elective conditions.

The patients will be taken to the endoscopy unit and hemodynamic monitoring will be applied. Vascular access will be opened and randomly divided into two groups as Group R (Restrictive, 2ml/kg 0.9% Sodium cloride-NaCl during colonoscopy) and Group L (Liberal 15ml/kg 0.9% NaCl during colonoscopy). For sedoanalgesia, Midazolam 0.02 mg/kg, Fentanyl 1 μg/kg, Ketamine 0.3 mg/kg will be administered intravenous (IV), followed by 10 mg additional doses of propofol until the Ramsay sedation score (RSS) is 3-4. All colonoscopy procedures will be performed by the same gastroenterologist.

During the colonoscopy procedure, patients will be given 3L/min oxygen with a face mask. Basal measurement values; heart rate, systolic arterial pressure, diastolic arterial pressure, mean arterial pressure, peripheral oxygen saturation (SpO2), respiratory rate and RSS will be recorded at regular intervals after sedation until the end of the colonoscopy attempt. Total midazolam, fentanyl, propofol, and ketamine doses, induction time, colonoscopy time, cecum intubation time, recovery time, and discharge time will be recorded. Possible hypoventilation, apnea, airway obstruction, hypotension, hypertension, arrhythmia, bradycardia, SpO2 falling below 95% and other side effects will be treated and recorded.

At the end of the procedure, the satisfaction of the gastroenterologist will be recorded. Patients with an RSS ≥2 will be admitted to the recovery unit, and patients with a postanesthetic discharge score of ≥9 will be sent home with an accompanying person. Recalls about the colonoscopy procedure by calling 24 hours after the procedure; Undesirable effects such as nausea, vomiting, pain, dizziness, drowsiness and satisfaction with the procedure will be questioned.

Expectations and scientific contributions This research may help to understand the effects of giving or not administering intravenous fluids (restrictive/liberal) prior to the procedure in patients undergoing elective colonoscopy under sedoanalgesia. It can provide hemodynamic stability, reduction in drug doses, reduction of side effects, rapid recovery and discharge, and reduction of costs.

ELIGIBILITY:
Inclusion Criteria:

1. Signing the informed consent form
2. Having irritable bowel disease, suspected colitis, unexplained iron deficiency and planning colonoscopy for screening
3. Between the ages of 18-65
4. According to the Physical Condition Classification of the American Society of Anesthesiologists, ASA I (a healthy person who does not cause normal systemic disorders, does not have a disease or systemic problem other than intestinal pathology) or ASA II (Person with mild systemic disorder due to a cause requiring intervention or another disease)

Exclusion Criteria:

1. Not signing the informed consent form
2. Not between the ages of 18-65
3. Having epileptic seizures
4. The use of drugs that affect the nervous system
5. Having a history of allergic reaction to study drugs
6. Long-term use of sedatives or sedatives
7. Receiving general anesthesia in the last 7 days
8. Having adrenocortical insufficiency (hormone deficiency)
9. Pregnancy
10. Having a psychiatric disorder
11. Having irritable bowel disease
12. Presence of nausea, vomiting or dizziness before the procedure
13. Being overweight
14. Having a bad general condition
15. Having had bowel surgery
16. Being in the risky patient group (>ASA II)
17. Alcohol addiction, inappropriate usage
18. Multiple biopsies during the procedure, unwanted bleeding, changes in the amount of fluid to be given

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of systolic blood pressure in restrictive and liberal patients in colonosopy under sedoanalgesia. | During colonoscopy
  Systolic blood pressure will be recoded.
Comparison of diastolic blood pressure in restrictive and liberal patients in colonosopy | During colonoscopy
  Diastolic blood pressure will be recoded.
Comparison of heart rate in restrictive and liberal patients in colonosopy | During colonoscopy
  Heart rate will be recoded.
Comparison of spO2 in restrictive and liberal patients in colonosopy | During colonoscopy
  spO2 will be recoded.
Comparison of procedure times in restrictive and liberal patients in colonosopy | During colonoscopy
  Procedure times will be recoded.
Comparison of total anaesthetic doses in restrictive and liberal patients in colonosopy | During colonoscopy
  Total anaesthetic doses will be recoded.
Comparison of nose and vomiting and other effects in restrictive and liberal patients in colonosopy | 24 hours
  Side effects will be recorded
Comparison of sedation levels in restrictive and liberal patients in colonosopy | 24 hours
  Ramsey and modified post anaesthetic discharge score level will be recorded.

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours
  Patient satisfaction will be assessed using a three point scale (satisfactory, moderate, not satisfactory) at the end of the procedure and after 24 hours via phone call. The patients will also be asked whether they have experienced any side effects (nausea, vomiting, abdominal pain, hallucination, double vision, etc.), and whether they would like to have the same sedoanalgesia procedure in the future colonoscopy procedures or not.
Gastroenterologist satisfaction | 24 hours
  At the end of the procedure, the gastroenterologist's opinion about our sedoanalgesia method will be evaluated.using a three point scale (satisfactory, moderate or unsatisfactory)..

CONTACTS AND LOCATIONS:
Overall Officials: Yonca Özvardar Pekcan, Principal Investigator — Baskent University
Locations (1):
- Baskent University Zubeyde Hanim Practice and Research Center, Izmir, Karşıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trummel JM, Chandrasekhara V, Kochman ML. Anesthesia for Colonoscopy and Lower Endoscopic Procedures. Anesthesiol Clin. 2017 Dec;35(4):679-686. doi: 10.1016/j.anclin.2017.08.007. PMID 29101957
- [Background] Tuncali B, Pekcan YO, Celebi A, Zeyneloglu P. Addition of low-dose ketamine to midazolam-fentanyl-propofol-based sedation for colonoscopy: a randomized, double-blind, controlled trial. J Clin Anesth. 2015 Jun;27(4):301-6. doi: 10.1016/j.jclinane.2015.03.017. Epub 2015 Mar 20. PMID 25801162
- [Background] das Neves JF, das Neves Araujo MM, de Paiva Araujo F, Ferreira CM, Duarte FB, Pace FH, Ornellas LC, Baron TH, Ferreira LE. Colonoscopy sedation: clinical trial comparing propofol and fentanyl with or without midazolam. Braz J Anesthesiol. 2016 May-Jun;66(3):231-6. doi: 10.1016/j.bjane.2014.09.014. Epub 2016 Mar 12. PMID 27108817
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Wexner SD, Beck DE, Baron TH, Fanelli RD, Hyman N, Shen B, Wasco KE; American Society of Colon and Rectal Surgeons; American Society for Gastrointestinal Endoscopy; Society of American Gastrointestinal and Endoscopic Surgeons. A consensus document on bowel preparation before colonoscopy: prepared by a task force from the American Society of Colon and Rectal Surgeons (ASCRS), the American Society for Gastrointestinal Endoscopy (ASGE), and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Gastrointest Endosc. 2006 Jun;63(7):894-909. doi: 10.1016/j.gie.2006.03.918. No abstract available. PMID 16733101
- [Background] 6. Indrakrishnan I and Varatharajah T. Management of Endoscopy Patients' Hydration Status during National Shortage of Intravenous Fluids. J Gastroenterol Liver Dis 2016; 1: 1001
- [Background] Leslie K, Allen M, Lee A, Clarke P. A randomized-controlled trial of high- or low-volume intravenous Plasma-Lyte((R)) to prevent hypotension during sedation for colonoscopy. Can J Anaesth. 2016 Aug;63(8):952-61. doi: 10.1007/s12630-016-0672-4. Epub 2016 May 18. PMID 27194403
- [Background] Leslie K, Tay T, Neo E. Intravenous fluid to prevent hypotension in patients undergoing elective colonoscopy. Anaesth Intensive Care. 2006 Jun;34(3):316-21. doi: 10.1177/0310057X0603400314. PMID 16802483
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468